CLINICAL TRIAL: NCT01896726
Title: The Effects of Multiple Doses of Baricitinib on the Pharmacokinetics of a Single Dose of an Oral Contraceptive in Healthy Female Subjects
Brief Title: A Study of Baricitinib and Birth Control Pills in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14601; I4V-MC-JAGD (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baricitinib + Microgynon (Experimental): Microgynon [30 micrograms (µg) ethinyl estradiol and 150 µg levonorgestrel] administered orally, once daily (QD), on Days 1 and 29. Baricitinib, 10 milligrams (mg), administered orally QD on Days 23 through 30.
  Interventions: Drug: Baricitinib; Drug: Microgynon

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
Drug: Microgynon — Administered orally

SUMMARY:
The main purpose of this study is to find out how the body absorbs and breaks down a common birth control pill called Microgynon when it is given with the study drug called baricitinib. Safety and the body's ability to tolerate baricitinib and Microgynon will also be studied. The study will last approximately 6 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females currently successfully using non-hormonal methods of contraception including tubular ligation, cervical vault cap, diaphragm, or non-hormonal coil with spermicide will be required in addition to use a second approved method of contraception for the duration of the study [that is (i.e.), a male sexual partner who agrees to use a male condom with spermicide; a sterile sexual partner; or abstinence (participants reporting abstinence who become sexually active while on the study must agree to use other additional barrier methods of contraception)]. The pregnancy test result must be negative at screening and at each check-in visit. Participants must have a regular menstrual cycle of approximately 28 days duration for at least 4 previous cycles prior to screening
* Postmenopausal females, or women not of child-bearing potential due to surgical sterilization (at least 3 months after surgical hysterectomy, or at least 3 months after bilateral oophorectomy or bilateral tubal occlusion with or without hysterectomy) confirmed by medical history, or menopause. Menopausal women include women with spontaneous amenorrhea for at least 12 months or amenorrhea not induced by a medical condition such as anorexia nervosa and/or not taking medications during that time of amenorrhea [example (e.g.), oral contraceptives (OCs), hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy]. Postmenopausal status should be confirmed by a serum follicle-stimulating hormone level at screening greater than 40 international units per liter (IU/L)
* Have a body mass index of 18 to 30 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Have a positive pregnancy test or are lactating
* Are currently enrolled in, have completed or discontinued within the last 90 days from a clinical trial involving a study drug; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are persons who have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received the study drug
* Have known allergies to baricitinib or Microgynon (containing ethinyl estradiol and levonorgestrel) or related compounds
* Have used or intend to use drugs or substances that are known to be inducers or inhibitors of cytochrome P450 3A (eg, St. John's wort, rifampin, ketoconazole) within 30 days prior to the first dose
* Have taken OCs within 3 months, implanted contraceptives within 6 months, injectable contraceptives within 12 months, or topical controlled delivery contraceptives (patch) or hormonal coils within 3 months prior to the study
* Have a history or presence of any thromboembolic disease, recurrent jaundice, acute or chronic liver disease, hormonally-induced migraines, undiagnosed vaginal bleeding, significant hyperlipidemia, and mammary, endometrial, or hepatic carcinoma (known or suspected)
* Smokes more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, fixed-sequence, 2-period study. Each participant received a single dose of Microgynon on Day 1 of Treatment Period 1. During Treatment Period 2, participants received baricitinib on Days 23 through 30 with coadministration of Microgynon on Day 29.
Groups:
- Baricitinib + Microgynon: Microgynon tablet [30 micrograms (µg) ethinyl estradiol and 150 µg levonorgestrel] administered orally, once daily (QD), on Days 1 and 29. 10 milligrams (mg) baricitinib tablet administered orally, QD, on Days 23 through 30.
Period: Treatment Period 1 (Days 1-22)
Arm/Group | Baricitinib + Microgynon
Started | 20
Received Microgynon | 20
Completed | 20
Not Completed | 0
Period: Treatment Period 2 (Days 23-31)
Arm/Group | Baricitinib + Microgynon
Started | 20
Received at Least 1 Dose of Baricitinib | 20
Received Microgynon | 18
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Baricitinib + Microgynon: Microgynon tablet (30 µg ethinyl estradiol and 150 µg levonorgestrel) administered orally, QD, on Days 1 and 29. 10 mg baricitinib tablet administered orally, QD, on Days 23 through 30.
Arm/Group | Baricitinib + Microgynon
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ethinyl Estradiol
Time Frame: Days 1 and 29: predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 and 48 hours post dose
Population: All enrolled participants who received study drug (Microgynon in Period 1 and at least 1 dose of baricitinib and Microgynon in Period 2) and had PK data to calculate Cmax of ethinyl estradiol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter (pg/mL)
Groups:
- Microgynon Alone: Microgynon tablet (30 µg ethinyl estradiol and 150 µg levonorgestrel) administered orally, QD, on Day 1
- Baricitinib + Microgynon: 10 mg baricitinib tablet administered orally, QD, on Days 23 through 30 with coadministration of Microgynon tablet (30 µg ethinyl estradiol and 150 µg levonorgestrel) administered orally, QD, on Day 29.
Arm/Group | Microgynon Alone | Baricitinib + Microgynon
Number analyzed (Participants) | 20 | 18
picograms/milliliter (pg/mL) | 63.8 (23) | 59.7 (24)

2. Primary Outcome: PK: Cmax of Levonorgestrel
Time Frame: Days 1 and 29: predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 and 48 hours post dose
Population: All enrolled participants who received study drug (Microgynon in Period 1 and at least 1 dose of baricitinib and Microgynon in Period 2) and had PK data to calculate Cmax of levonorgestrel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Microgynon Alone | Baricitinib + Microgynon
Number analyzed (Participants) | 20 | 18
pg/mL | 3390 (34) | 3340 (26)

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity [AUC(0-∞)] of Ethinyl Estradiol
Time Frame: Days 1 and 29: predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 and 48 hours post dose
Population: All enrolled participants who received study drug (Microgynon in Period 1 and at least 1 dose of baricitinib and Microgynon in Period 2) and had PK data to calculate AUC(0-∞) of ethinyl estradiol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hour/milliliter (pg*hr/mL)
Arm/Group | Microgynon Alone | Baricitinib + Microgynon
Number analyzed (Participants) | 20 | 18
picograms*hour/milliliter (pg*hr/mL) | 694 (24) | 697 (25)

4. Primary Outcome: PK: AUC(0-∞) of Levonorgestrel
Time Frame: Days 1 and 29: predose and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24 and 48 hours post dose
Population: All enrolled participants who received study drug (Microgynon in Period 1 and at least 1 dose of baricitinib and Microgynon in Period 2) and had PK data to calculate AUC(0-∞) of levonorgestrel.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Microgynon Alone | Baricitinib + Microgynon
Number analyzed (Participants) | 20 | 18
pg*hr/mL | 48200 (58) | 42400 (45)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 40).
Groups:
- Microgynon Alone: Microgynon tablet (30 µg ethinyl estradiol and 150 µg levonorgestrel) administered orally, QD, on Day 1.
  Adverse events are reported from baseline through predose on Day 23.
- Baricitinib: 10 mg baricitinib tablet administered orally, QD, on Days 23 through 28.
  Adverse events are reported from postdose on Day 23 through predose on Day 29.
- Baricitinib + Microgynon: 10 mg baricitinib tablet administered orally, QD, on Days 29 through 30 with coadministration of Microgynon tablet (30 µg ethinyl estradiol and 150 µg levonorgestrel) administered orally, QD, on Day 29.
  Adverse events are reported from postdose on Day 29 up to Day 40.
Arm/Group | Microgynon Alone | Baricitinib | Baricitinib + Microgynon
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/18
Other Adverse Events (participants affected / at risk) | 3/20 | 4/20 | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microgynon Alone (N=20) | Baricitinib (N=20) | Baricitinib + Microgynon (N=18)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microgynon Alone (N=20) | Baricitinib (N=20) | Baricitinib + Microgynon (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days